CLINICAL TRIAL: NCT01044901
Title: Cardiovascular Complications of Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16653A
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Cardiac magnetic resonance imaging; Coronary Disease; Pulmonary Hypertension
MeSH Terms: conditions — Anemia, Sickle Cell; Coronary Disease; Hypertension, Pulmonary | interventions — Magnetic Resonance Spectroscopy; Manometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will study blood samples for chemicals related to sickle cell and heart and lung disease, and will be evaluating DNA for purposes of the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with Sickle Cell Disease (SCD): 38 clinically stable black patients with Sickle Cell Disease (SCD) (including individuals with hemoglobin SS, SC, and β-thalassemia demonstrated by high-performance liquid chromatographic separation or gel electrophoresis).
  Interventions: Procedure: MRI, Transthoracic Echocardiography, tonometry, EKG
- Healthy Volunteers: 13 healthy control subjects were frequency matched to patients with SCD on age, sex, and race.
  Interventions: Procedure: MRI, Transthoracic Echocardiography, tonometry, EKG

INTERVENTIONS:
Procedure: MRI, Transthoracic Echocardiography, tonometry, EKG — Unless contraindicated, subjects will receive Regadenoson and Gadolinium contrast agent during the Cardiac magnetic resonance. The tonometer, EKG, and echo are non-invasive procedures.
  Other Names: electrocardiography; Cardiac magnetic resonance; Doppler trans-thoracic echocardiography

SUMMARY:
In this research study, we are using heart imaging exams and blood testing, in order to gain an improved understanding of the pulmonary (lung) hypertension and cardiovascular (heart) complications that often occur in sickle cell patients. Information gathered from the healthy volunteers that participate in this study will be compared to information from the sickle cell patients in this study in order to help further our understanding.

DETAILED DESCRIPTION:
Cardiac magnetic resonance (CMR) has gained increasing clinical application in cardiopulmonary diseases. Due to its 3-dimensional nature, CMR is considered the gold-standard for quantifying left and right ventricular systolic function and size. Additionally, its high tissue contrast allows for a detailed characterization of myocardial tissue. Specifically, the use of techniques such as late gadolinium enhancement can be used to detect the presence of tiny amounts of myocardial scar. Other techniques have been shown to correlate strongly with myocardial iron content. Just as importantly, CMR perfusion imaging can accurately quantify myocardial blood flow and can provide tremendous insight into the function of the microcirculation. CMR's high spatial and temporal resolution, its 3-dimensional approach, its ability to characterize the tissue, and its ability to evaluate the micro- and macro-circulation make it a comprehensive technique for the evaluation of heart disease. Recently, one CMR study has already shown the presence of cardiac microvascular disease in a subset of adult sickle cell disease (SCD) patients in the absence of infarcted myocardium, myocardial iron overload, or coronary artery disease, increasing the evidence for the contribution of left heart disease to pulmonary hypertension (PH) development in these patients; unfortunately, strong conclusions could not be made because the study was underpowered. Thus, this proposal will leverage the advantages offered by CMR to better characterize and detect the PH and cardiopulmonary subphenotypes in the SCD patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18+
* Patients who were diagnosed with SCD confirmed by high-pressure liquid chromatography or hemoglobin electrophoresis will be eligible for the study
* Only patients in stable condition will be included
* Patients receiving transfusions will not be excluded

Exclusion Criteria:

* Patients with vaso-occlusive crises or an episode of acute chest syndrome within the previous four weeks (after 4 weeks have passed, the patients may be re-evaluated for eligibility)
* Patients with high degree heart block; active, hemodynamically significant, ventricular arrhythmias; unstable coronary syndromes; history of myocardial infarction within 1 month of the study.
* Contraindications to gadolinium-enhanced magnetic resonance examination such as severe claustrophobia, Pacemaker, defibrillators, cerebral aneurysm clips, or neurostimulator.
* Pregnancy
* Patients with sinus node dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from clinics at the University of Chicago as well as from the community via flyers posted at the University of Chicago and a web site posted on the University of Chicago Medical Center web site.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2009-03; Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit R Patel, M.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Desai AA, Patel AR, Ahmad H, Groth JV, Thiruvoipati T, Turner K, Yodwut C, Czobor P, Artz N, Machado RF, Garcia JGN, Lang RM. Mechanistic insights and characterization of sickle cell disease-associated cardiomyopathy. Circ Cardiovasc Imaging. 2014 May;7(3):430-437. doi: 10.1161/CIRCIMAGING.113.001420. Epub 2014 Mar 27. PMID 24676783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Started | 38 | 13
Completed | 38 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers | Total
Number analyzed (Participants) | 38 | 13 | 51
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 32 [27 to 38] | 25 [23 to 43] | 29 [23 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 8 | 29
  Male | 17 | 5 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 13 | 51
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Surface Area [Median (Inter-Quartile Range); unit: m^2] | 2.0 [1.7 to 2.1] | 1.8 [1.7 to 1.9] | 2.0 [1.7 to 2.1]

OUTCOME MEASURES:

1. Primary Outcome: MRI Parameter - LVEDVi, mL/cm2 (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: Comprehensively and quantitatively characterized the cardiopulmonary complications of SCD and gained an improved understanding of the pathophysiology of pulmonary hypertension and diastolic dysfunction in patients with Sickle Cell Disease.
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: mL/cm2
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
mL/cm2 | 124.0 (26.8) | 78.7 (11.9)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; Primary outcome was presented at baseline as mean +/- standard deviation based upon the Shapiro-Wilks test of normality, and then analyzed with a Student t-test; Test type: Other; p = 0.0039, t-test, 2 sided — P-values are not adjusted for multiple comparisons. Tests were two-tailed, considered statistically significant with a p-value <0.05

2. Primary Outcome: MRI Parameter - LVESVi, mL/cm2 - (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Median (Inter-Quartile Range); unit: mL/cm2
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
mL/cm2 | 47 [39 to 62] | 31 [24 to 37]
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; Primary outcome was presented at baseline as median (interquartile range) based upon the Shapiro-Wilks test of normality, and then analyzed with a Wilcoxon (Mann-Whitney test); Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: MRI Parameter - LV Mass Index, g/cm2, (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
g/cm2 | 77.2 (19.2) | 51.6 (13.6)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0137, t-test, 2 sided; P-values are not adjusted for multiple comparisons. Tests were two-tailed, considered statistically significant with a p-value <0.05

4. Primary Outcome: MRI Parameter - RVEDVi, mL/cm2, (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: mL/cm2
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
mL/cm2 | 126.4 (27.7) | 83.0 (13.7)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0039, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

5. Primary Outcome: MRI Parameter - RVESVi, mL/cm2, (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: mL/cm2
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
mL/cm2 | 56.3 (17.1) | 37.8 (7.2)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.16, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

6. Primary Outcome: MRI Parameter - LAi, mL/cm2, (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: mL/cm2
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
mL/cm2 | 64.8 (16.2) | 41.1 (9.1)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0039, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

7. Primary Outcome: MRI Parameter - RAi, mL/cm2, (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Median (Inter-Quartile Range); unit: mL/cm2
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
mL/cm2 | 76 [66 to 86] | 52 [48 to 56]
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; Primary outcome was presented at baseline as median (interquartile range) based upon the Shapiro-Wilks test of normality, and then analyzed with a Wilcoxon (Mann-Whitney) test; Test type: Other; p = 0.0011, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

8. Primary Outcome: MRI Parameter - LVEF, %, (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Median (Inter-Quartile Range); unit: percentage of ejection fraction
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
percentage of ejection fraction | 58 [55 to 62] | 64 [56 to 67]
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.10, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

9. Primary Outcome: MRI Parameter - RVEF, %, (Measured Using Method of Disks, Controls Serve as Normal Ranges)
Description: as for outcome 1
Time Frame: Parameter at baseline.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
percentage of ejection fraction | 56.1 (6.4) | 55.4 (2.7)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.48, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

10. Primary Outcome: MRI Parameter - Late Gadolinium Enhancement, Performed Via Visual Inspection, Normally None Should be Present
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Population: Some parameters were unable to be collected from patients with Sickle Cell Disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 32 | 13
Participants | 8 | 0
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; Primary outcome was presented as frequencies and percentages, and then analyzed with a Fisher exact test; Test type: Other; p = 0.08, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

11. Primary Outcome: MRI Parameter - Myocardial T2-star, ms, Performed Using Decay Curves (Normal >20ms)
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
ms | 41.6 (13.4) | 38.4 (14.4)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.91, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

12. Primary Outcome: MRI Parameter - Hepatic T2-star, ms, Performed Using Decay Curves, Normal >18ms
Description: as for outcome 1
Time Frame: Parameter at baseline.
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
ms | 10 [5 to 27] | 30 [24 to 38]
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0038, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

13. Primary Outcome: MRI Parameter - Myocardial Perfusion Reserve Index, Measured Using Upslope Technique. Control Subjects Available for Normal Ranges
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
index | 1.4 (0.3) | 1.87 (0.37)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.034, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

14. Primary Outcome: MRI Parameter - Diastolic Dysfunction, Determined According to American Society of Echocardiography Guidelines
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Population: The measure was unable to be measured for some patients with Sickle Cell Disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 35 | 13
Participants | 10 | 1
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; Primary outcome was presented was as frequencies and percentages, and then analyzed with a Fisher exact test; Test type: Other; p = 0.25, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

15. Primary Outcome: MRI Parameter - Lateral E/e', Measured Using Doppler Echo. Controls Available as Normal Ranges
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
ratio | 7.2 [5.9 to 9.8] | 6.0 [5.1 to 6.7]
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.0288, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

16. Primary Outcome: MRI Parameter - Augmentation Pressure, See Controls for Normal Ranges
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Median (Inter-Quartile Range); unit: percentage of the pulse pressure
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
percentage of the pulse pressure | 9.0 [4.5 to 16.8] | 2.0 [0.3 to 14.1]
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.14, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

17. Primary Outcome: MRI Parameter - Augmentation Index, See Control Subjects for Normal Ranges
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
index | 23.6 (16.2) | 12.5 (20.4)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.13, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

18. Primary Outcome: MRI Parameter - Systemic Systolic Blood Pressure
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
mmHg | 122.3 (21.7) | 132 (17.6)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.81, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

19. Primary Outcome: MRI Parameter - Systemic Diastolic Blood Pressure, mm Hg
Description: as for outcome 1
Time Frame: Parameter measured at baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 38 | 13
mmHg | 68.3 (18.1) | 74.9 (16.3)
Statistical Analysis 1: Comparison: Subjects With Sickle Cell Disease (SCD) vs Healthy Volunteers; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.30, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

20. Secondary Outcome: Genome-Wide Gene Expression and Targeted Genetic Polymorphisms in SCD Patients Linked to a Quantitative Noninvasive-based PH Phenotype.
Description: To detect genome-wide gene expression and targeted genetic polymorphisms in SCD patients linked to a quantitative noninvasive-based PH phenotype.
Time Frame: median follow up 3 years
Population: All efforts were taken to gather all possible data but none were obtained for this Outcome Measure.
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 3 years.
Arm/Group | Subjects With Sickle Cell Disease (SCD) | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 3/38 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/13
Other Adverse Events (participants affected / at risk) | 0/38 | 0/13

LIMITATIONS AND CAVEATS:
Due to small sample size, caution should be considered in applying these results to all patients with SCD, in particular to those with genotypes outside of hemoglobin and those with a recent or ongoing crisis. Not all patients had evaluable data sets for all of the cardiovascular tests, due to inadequate venous access, frequently encountered in patients with SCD. Finally, our follow-up period is currently too short to make meaningful comments on outcomes such as mortality and functional status.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2009-03-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT01044901/Prot_SAP_ICF_001.pdf